CLINICAL TRIAL: NCT03988920
Title: A Long-Term, Open Label Study to Evaluate the Ability of Tenapanor Alone or in Combination With Sevelamer to Treat to Goal Serum Phosphorus in Patients With End-Stage Kidney Disease on Dialysis (NORMALIZE)
Brief Title: A Long-Term Study of Tenapanor Alone or in Combination With Sevelamer in Patients With CKD on Dialysis and HP
Acronym: NORMALIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEN-02-401
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Hyperphosphatemia; End Stage Renal Disease
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — tenapanor; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenapanor w/Sevelamer (Experimental): Tenapanor will be administered QD or BID and sevelamer can be added to achieve desired serum phosphorus level
  Interventions: Drug: Tenapanor; Drug: Sevelamer Carbonate
- Sevelamer w/Tenapanor (Experimental): Sevelamer will be administered QD, BID or TID and tenapanor will be added to achieve desired serum phosphorus level and sevelamer dose will be decreased as needed
  Interventions: Drug: Tenapanor; Drug: Sevelamer Carbonate

INTERVENTIONS:
Drug: Tenapanor — NHE3 Inhibitor
Drug: Sevelamer Carbonate — Phosphate binder

SUMMARY:
The study is designed to evaluate the ability of tenapanor alone or in combination with sevelamer to achieve serum phosphorus concentration (sP) within the population reference range (sP >2.5 and ≤4.5 mg/dL) in patients with end-stage renal disease (ESRD) on dialysis with hyperphosphatemia (>4.5 mg/dL).

DETAILED DESCRIPTION:
Patients who complete the TEN-02-301 study (PHREEDOM) may be eligible to enroll into TEN-02-401 (NORMALIZE).

Patients from the TEN-02-301 tenapanor arm will either receive only tenapanor or be given sevelamer in addition to tenapanor based on their sP. Patients from the TEN-02-301 sevelamer arm will be given tenapanor in addition to their sevelamer dose and the sevelamer dose will then be adjusted based on their sP following a protocol-specified dose titration schedule. Patients will be monitored for safety and efficacy with in-office and telephone visits for up to an additional 18 months.

Laboratory assessments will be measured at every visit (Weeks 1, 2, 3, 4, 6 and 8 and Months 3, 6, 9, 12, 15 and 18) using a central laboratory.

Safety assessments will be performed during the study and will include physical examinations, vital signs (blood pressure and pulse), body weights, clinical laboratory evaluations, 12-lead electrocardiograms (ECGs), and adverse event (AE) monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Must complete TEN-02-301 (PHREEDOM)

Exclusion Criteria:

1. Schedlued for kidney transplant
2. Life expectancy <12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, PhD, Study Director — Ardelyx
Locations (1):
- Ardelyx Site #509, Houston, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sprague SM, Weiner DE, Tietjen DP, Pergola PE, Fishbane S, Block GA, Silva AL, Fadem SZ, Lynn RI, Fadda G, Pagliaro L, Zhao S, Edelstein S, Spiegel DM, Rosenbaum DP. Tenapanor as Therapy for Hyperphosphatemia in Maintenance Dialysis Patients: Results from the OPTIMIZE Study. Kidney360. 2024 May 1;5(5):732-742. doi: 10.34067/KID.0000000000000387. Epub 2024 Feb 7. PMID 38323855
- [Derived] Silva AL, Chertow GM, Hernandez GT, Lynn RI, Tietjen DP, Rosenbaum DP, Yang Y, Edelstein S. Tenapanor Improves Long-Term Control of Hyperphosphatemia in Patients Receiving Maintenance Dialysis: the NORMALIZE Study. Kidney360. 2023 Nov 1;4(11):1580-1589. doi: 10.34067/KID.0000000000000280. Epub 2023 Oct 19. PMID 37853560

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenapanor w/Sevelamer | Sevelamer w/Tenapanor
Started | 111 | 61
Completed | 89 | 35
Not Completed | 22 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenapanor w/Sevelamer | Sevelamer w/Tenapanor | Total
Number analyzed (Participants) | 111 | 61 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.97 (12.146) | 58.48 (14.028) | 56.85 (12.861)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 17 | 63
  Male | 65 | 44 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 20 | 51
  Not Hispanic or Latino | 80 | 41 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 0 | 7
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 59 | 27 | 86
  White | 44 | 31 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 61 | 172
Region of Enrollment [Number; unit: participants]
  United States | 111 | 61 | 172
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.90 (7.360) | 29.33 (7.472) | 30.98 (7.480)

OUTCOME MEASURES:

1. Primary Outcome: Achieving Normal Serum Phosphorus Level
Description: Proportion of patients with serum phosphorus between 2.5 and 4.5 mg/dL
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tenapanor w/Sevelamer | Sevelamer w/Tenapanor
Number analyzed (Participants) | 111 | 60
Participants | 36 | 21
Statistical Analysis 1: Comparison: Tenapanor w/Sevelamer vs Sevelamer w/Tenapanor; Test type: Superiority; p = 0.7439, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.9

2. Secondary Outcome: Change in Serum Phosphorus (s-P) From TEN-02-301 (Parent Study) Baseline
Description: The change from the baseline s-P from the parent study until the endpoint visit which was up to 2.5 years after the baseline
Time Frame: up to 2.5 years
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tenapanor w/Sevelamer | Sevelamer w/Tenapanor
Number analyzed (Participants) | 111 | 60
mg/dL | -2.00 (2.248) | -1.91 (1.982)

3. Secondary Outcome: Change From Baseline in Serum Phosphorus (of Extension Study; TEN-02-401) to Endpoint Visit
Description: Baseline upon enrollment in the 18-month long-term extension study
Time Frame: up to 18 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tenapanor w/Sevelamer | Sevelamer w/Tenapanor
Number analyzed (Participants) | 111 | 60
mg/dL | -0.47 (2.084) | -0.57 (2.422)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Groups:
- Sevelamer w/Tenapanor: Tenapanor will be added and sevelamer dose will be decreased immediately after enrollment to achieve desired phosphorus level.
  Tenapanor: NHE3 Inhibitor
  Sevelamer Carbonate: Phosphate binder
Arm/Group | Tenapanor w/Sevelamer | Sevelamer w/Tenapanor
All-Cause Mortality (participants affected / at risk) | 5/111 | 4/61
Serious Adverse Events (participants affected / at risk) | 56/111 | 22/61
Other Adverse Events (participants affected / at risk) | 91/111 | 52/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenapanor w/Sevelamer (N=111) | Sevelamer w/Tenapanor (N=61)
COVID-19 (Infections and infestations) | 6 | 1
COVD-19 pnuemonia (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 3 | 1
Celulitis (Infections and infestations) | 2 | 3
Sepsis (Infections and infestations) | 3 | 2
Acute Myocardial Infarction (Cardiac disorders) | 3 | 2
Cardiac Failure Congestive (Cardiac disorders) | 2 | 2
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 1
Arteriovenous Fistula Aneurysm (Injury, poisoning and procedural complications) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertensive Urgency (Vascular disorders) | 2 | 0
Haemorrhage Intracranial (Nervous system disorders) | 2 | 0
Ischaemic Stroke (Nervous system disorders) | 2 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical Device Site Joint Infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenapanor w/Sevelamer (N=111) | Sevelamer w/Tenapanor (N=61)
Diarrhoea (Gastrointestinal disorders) | 11 | 27
COVID-19 (Infections and infestations) | 8 | 4
Cellulitis (Infections and infestations) | 7 | 3
Nasopharyngitis (Infections and infestations) | 9 | 1
Pneumonia (Infections and infestations) | 5 | 4
Sepsis (Infections and infestations) | 6 | 2
Nausea (Gastrointestinal disorders) | 8 | 2
Vomiting (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 3 | 4
Fall (Injury, poisoning and procedural complications) | 9 | 6
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 7 | 1
Hypertension (Vascular disorders) | 7 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 3
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Troponin Increased (Investigations) | 1 | 4
Hypotension (Vascular disorders) | 8 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03988920/Prot_SAP_000.pdf